CLINICAL TRIAL: NCT03198910
Title: Efficacy of Medical Therapy for Pulmonary Arterial and Inoperable Chronic Thromboembolic Pulmonary Hypertension in a Real Life Setting
Brief Title: Retrospective Data Analysis of Data From the Zurich PH Registry
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2016-00786
Record Dates: First submitted 2017-06-20; First posted 2017-06-26 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Artery Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary arterial hypertension
- Chronic thromboembolic pulmonary hypertension

SUMMARY:
The collected data from the Zurich Registry for pulmonary Hypertension (PH) are evaluated in a retrospective analysis. This study examines the number of patients and their exact diagnoses who are treated at the University Hospital of Zurich and potentially other participating in the Zurich Registry. Other demographic parameters such as age, gender and body-mass-index are also part of the evaluation. Furthermore, the analysis will focus on the newest guidelines on PH. Therefore, it will be checked how many patients would fulfill the therapeutic goals in terms of New York Heart Classification (NYHA), 6-minute walk distance, sign of right heart failure and N-terminal pro-brain-natriuretic peptide(NTproBNP). Additionally, the study examines on how the patients are treated. Despite the different kind of Drugs, the focus lies on the combination therapy (single, double, triple) and the impact the therapy had on the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary arterial hypertension (PAH)
* Patients with chronic thromboembolic pulmonary hypertension (CTEPH)
* All prevalent patients (diagnosed >12 month ago) with PAH or distal CTEPH who had a consultation at the PH centre in Zurich between November 2015 and November 2016)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAH and CTEPH patients diagnosed with a right heart catheter
Sampling Method: Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in NYHA/WHO functional class | Baseline, 3 months, 6 months, 1 year
  Change of the functional class over time in relation to given vasodilator treatment
Change in 6 minute walk distance | Baseline, 3 months, 6 months, 1 year
  Change of the 6 minute walk distance over time in relation to given vasodilator treatment
Change in NT-proBNP | Baseline, 3 months, 6 months, 1 year
  Change of the 6 minute walk distance over time in relation to given vasodilator treatment

SECONDARY OUTCOMES:
Percentage of patients that are in NYHA/WHO functional class <= II | Baseline, 3 months, 6 months, 1 year
  Percentage of patients that are in NYHA/WHO functional class <= II will be assessed at respective timepoints
Percentage of patients with a 6 minute walk distance > 440m | Baseline, 3 months, 6 months, 1 year
  Percentage of patients with a 6 minute walk distance > 440m will be assessed at respective timepoints
Percentage of patients with a NT-proBNP < 300 ng/l | Baseline, 3 months, 6 months, 1 year
  Percentage of patients with a NT-proBNP < 300 ng/l will be assessed at respective timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No